CLINICAL TRIAL: NCT06131164
Title: Effects Of Breathing Exercises On Cardiorespiratory Parameters In Subjects With Forward Head Posture
Brief Title: Breathing Exercises Effects on Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0332
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Forward Head Posture
Keywords: Forward Head Posture; Diaphragmatic breathing exercise; Thoracic Extension Exercise; Cardiorespiratory parameters; Craniovertebral Angle

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic Breathing Exercise Group (Experimental): This group will perform baseline treatment along with balloon breathing exercises also known as diaphragmatic breathing exercise for pulmonary function improvement and FHP Diaphragmatic breathing is done slowly and deeply through nose with minimum usage of chest movement. Only diaphragm is used for breathing in supine lying position with one hand placed on chest and other hand is placed on abdomen. Focus should be on the contraction of diaphragm that can be checked by hand placed on abdomen while there is as little movement in chest as possible which is also checked by hand placed on chest. Inhalation and exhalation should be for 6 second approximately. Each exercise session consist of 4 sets and each set has 4 complete breathing breaks. Will be done 2 times a day and 3 times per week for total of 8 weeks.
  Interventions: Other: Diaphragmatic Breathing Exercise Group
- Thoracic Extension Exercise Group (Active Comparator): This group along with baseline treatment will do Thoracic Extension Exercises (TEE) for FHP and Pulmonary function improvements. This is done in 3 steps. The restricted upper thoracic area is placed on foam roller with subject lying supine with knees flexed, buttock slightly lifted up from the floor and crossed hands on the chest. Roll the foam roller slightly up and down. Swiss ball is place in front of the subject who is sitting with knees flexed and then the ball is pushed slightly forward with both hands placed on it. While lying prone lift up and then pushing down the upper body while the upper body is supported by elbows places just below shoulders. All these steps will be followed by 2 sets of 15 repetitions and holding 10 sec for each repetition.
  Interventions: Other: Thoracic Extension Exercise Group

INTERVENTIONS:
Other: Diaphragmatic Breathing Exercise Group — The subjects in this group will perform Diaphragmatic Breathing Exercise Group
  Arms: Diaphragmatic Breathing Exercise Group
Other: Thoracic Extension Exercise Group — The subjects in this group will perform Thoracic Extension Exercise Group
  Arms: Thoracic Extension Exercise Group

SUMMARY:
The main objective of this study is to find the effects of breathing exercises on cardiorespiratory parameters in subjects with forward head posture. This will be a Randomized Clinical Trial study with two different breathing exercises which include Diaphragmatic Breathing Exercise (DBE) for Treatment group A individuals and Thoracic Extension Exercise (TEE) for Treatment Group B individuals will be performed along with ergometric advices. Each exercise session will be done three times per week for total over a period of 12 weeks. Outcomes will be measured at baseline, 6th and 12th week with photogrammetry method for craniovertebral angle (CVA) and spirometer for pulmonary function test values (PFTs).

DETAILED DESCRIPTION:
The Forward Head Posture (FHP)is the poor posture alignment of the body in which the craniovertebral angle is <50 degrees. This FHP causes the deep cervical flexors to become weak and excessive use of the sternocleidomastoid and anterior scalene muscle leads towards compromised respiratory functions. The diaphragm mobility is also reduced which effect the lung volume and capacities.

FHP is due to weak deep neck flexor muscles which are compensated by the over-activity of sternocleidomastoid and scalene muscle. This in turn leads to many musculoskeletal changes like muscular imbalance, changes in stress-strain curve due to over activity of cervical spine. FHP can badly effect thoracic expansion and alveolar ventilation which can reduce vital capacity, reduce lung volumes and lung capacities thus leading towards respiratory function weakening.

Prolonged FHP not only affect the muscles but also involve ligaments of the cervical and upper thoracic spine which cause the respiratory disorders and the end result of these changes shows that 83% of individuals with this forward head posture had altered breathing pattern. This shows that there is strong relation between cervical posture and respiratory parameters.

The respiratory function is usually affected by any change in muscle activity which is caused by pain in neck flexors or extensors and their reduced activity which causes changes in vicious circle of the neck. For improvements in such forward head posture and its related problems many therapeutic and rehabilitative techniques have been used such as Kinesio tapping, myofascial release, and Mckenzie exercises.All of these showed positive impact in improving the forward head posture and reducing impairments. Some of the previous exercises mentioned showed the positive combined effects of breathing exercises and therapeutic exercises

ELIGIBILITY:
Inclusion Criteria:

* Both Males and Females are included
* Age group: Middle age adult from 30 to 45 years are included
* Individuals with forward head posture and Craniovertebral Angle <50o

Exclusion Criteria:

* Previous history of neck or back surgery or neurological signs
* Psoriatic arthritis or rheumatoid arthritis
* Currently using muscle relaxation medication
* Cervical fracture, trauma or tumor
* Unstable cardiac condition
* Undergone any thoracic or abdominal surgery

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Photogrammetry Method for Forward Head Posture Assessment | Baseline; 6th Week; 12th Week
  Photogrammetry is a reliable and accurate tool for measurement of angles. It is used to measure the FHP through measurement of Craniovertebral angle (CVA) measurement. CVA is the inner angle between the horizontal line drawn from C7 spinous process to the midpoint of the tragus. As the higher the CVA the higher the FHP. All measurements are done after taking a photograph via digital camera in lateral-view in standing position
Spirometry for Pulmonary Function Test FEV1 | Baseline; 6th Week; 12th Week
  Spirometry method is use to measure pulmonary functions by assessing the lung volumes and capacities. As these pulmonary values will changed after FHP as the mobility of cervical spine and diaphragm are compromised. Spirometry is a cost effect, environment friendly, noninvasive and sensitive tool which can easily help in assessment of pulmonary function
Spirometry for Pulmonary Function Test FVC | Baseline; 6th Week; 12th Week
  Spirometry method is use to measure pulmonary functions by assessing the lung volumes and capacities. As these pulmonary values will changed after FHP as the mobility of cervical spine and diaphragm are compromised. Spirometry is a cost effect, environment friendly, noninvasive and sensitive tool which can easily help in assessment of pulmonary function
Spirometry for Pulmonary Function Test FEV1/FVC ratio | Baseline; 6th Week; 12th Week
  Spirometry method is use to measure pulmonary functions by assessing the lung volumes and capacities. As these pulmonary values will changed after FHP as the mobility of cervical spine and diaphragm are compromised. Spirometry is a cost effect, environment friendly, noninvasive and sensitive tool which can easily help in assessment of pulmonary function

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No